CLINICAL TRIAL: NCT02515175
Title: A Randomized, Double-Blind Study to Evaluate a New Formulation of GEN-003 in Subjects With Genital HSV-2 Infection
Brief Title: Evaluating New Formulation of Therapeutic HSV-2 Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genocea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GEN-003-003
Record Dates: First submitted 2015-07-31; First posted 2015-08-04 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Genital Herpes Simplex Type 2
Keywords: HSV; Herpes; Genital Herpes; Vaccine
MeSH Terms: conditions — Herpes Simplex; Herpes Genitalis | interventions — M2 protein, Influenza A virus; Adjuvants, Pharmaceutic; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GEN-003 60ug / Matrix-M2 50ug (Experimental): GEN-003/M2 (60 ug of each antigen) with Matrix-M2 adjuvant (50ug), administered as a 0.5mL intramuscular (IM) injection
  Interventions: Biological: Matrix-M2; Biological: GEN-003
- GEN-003 60ug / Matrix-M2 75ug (Experimental): GEN-003/M2 (60 ug of each antigen) with Matrix-M2 adjuvant (75ug), administered as a 0.5mL intramuscular (IM) injection
  Interventions: Biological: Matrix-M2; Biological: GEN-003
- Placebo (Placebo Comparator): 0.9% Normal Saline administered as a 0.5 mL intramuscular (IM) injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Matrix-M2 — Matrix-M2 is derived from fractionated Quillaja saponins, phosphatidylcholine, and cholesterol.
  Other Names: Adjuvant
  Arms: GEN-003 60ug / Matrix-M2 50ug; GEN-003 60ug / Matrix-M2 75ug
Biological: GEN-003 — HSV-2 protein subunit vaccine consisting of 2 recombinant T cell antigens: internal fragment of the immediate early (IE) protein ICP and glycoprotein D
  Other Names: HSV Therapeutic Vaccine
  Arms: GEN-003 60ug / Matrix-M2 50ug; GEN-003 60ug / Matrix-M2 75ug
Drug: Placebo — 0.9% Normal Saline
  Other Names: 0.9% Normal Saline
  Arms: Placebo

SUMMARY:
This study evaluates the reduction in viral shedding after vaccination with a new formulation of GEN-003 in subjects with genital HSV-2 infection. Two-thirds of the participants will receive GEN-003, one-third will receive placebo.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled clinical trial of a new formulation of GEN-003 for treatment of HSV-2 genital infection.

Eligible subjects will enter a baseline period to collect anogenital swabs for 28 consecutive days prior to randomization. Each subject will receive up to 3 doses at 21 day intervals then complete a second set of anogenital swabs for 28 consecutive days after the third dose. Each subject will be followed for one year after the third dose.

ELIGIBILITY:
Inclusion Criteria

* A history of at least 3 and no more than 9 reported clinical occurrences in the prior 12 months, or, if currently on suppressive antiviral therapy, a history of at least 3 and no more than 9 reported clinical occurrences in the 12 months prior to initiation of antiviral suppressive therapy
* Diagnosis of genital HSV-2 infection for > 1 year
* Willing and able to provide written informed consent
* Willing to perform and comply with all study procedures including attending clinic visits as scheduled and completion of an electronic lesion report form
* Willing to not use suppressive antiviral therapy from 14 days prior to starting the study and for the duration of the study
* Men and women must be willing to practice a highly effective method of contraception that may include, but is not limited to, abstinence, sex only with persons of the same sex, monogamous relationship with vasectomized partner, vasectomy, tubal ligation, hysterectomy, licensed hormonal methods, intrauterine device, or barrier method (e.g., condom, diaphragm) with spermicide for 28 days before and 90 days after receiving the Study Drug

Exclusion Criteria

* On suppressive antiviral therapy within 14 days of starting the study
* Use of topical steroids or antiviral medication in the anogenital region within 14 days of starting the study and during study
* Use of tenofovir, lysine, or other medication or supplement known or purported to affect HSV outbreak frequency or intensity within 14 days of starting the study
* History of any form of ocular HSV infection, HSV-related erythema multiforme, or herpes meningitis or encephalitis
* Immunocompromised individuals
* Use of corticosteroids within 30 days of starting the study and during the study or other immunosuppressive agents
* Presence or history of autoimmune disease regardless of current treatment
* Current infection with HIV or hepatitis B or C virus
* History of hypersensitivity to any component of the vaccine
* Prior receipt of GEN-003 or another vaccine containing HSV-2 antigens
* Receipt of any investigational product within 30 days prior to Dose 1
* Receipt of blood products within 90 days prior to Dose 1
* Planned use of any vaccine over the course of the study
* Pregnant or nursing women
* History of drug or alcohol abuse
* Other active, uncontrolled comorbidities

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2015-11; Primary Completion 2016-07 (Actual); Study Completion 2017-05-25 (Actual)

PRIMARY OUTCOMES:
Change in HSV-2 viral shedding rate | baseline (Days -28 to Day 1) and after vaccination (Days 43 to 71)

SECONDARY OUTCOMES:
Immunogenicity measured by humoral (antibody) responses to vaccine antigens | 13 weeks
Impact on clinical HSV-2 disease based on time to first recurrence | 64 weeks
Number of patients with adverse events as a measure of safety and tolerability | 64 weeks
Reduction in HSV-2 viral shedding rate | After vaccination (6 Months and 12 Months)
Impact on clinical HSV-2 disease based on lesion rate | 64 weeks
Impact on clinical HSV-2 disease based on percent recurrence-free | 64 weeks

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Medical Center for Clinical Research, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - The Fenway Institute, Boston, Massachusetts
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Childrens Hospital, Cincinnati, Ohio
  - Tekton Research, Austin, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bernstein DI, Flechtner JB, McNeil LK, Heineman T, Oliphant T, Tasker S, Wald A, Hetherington S; Genocea study group. Therapeutic HSV-2 vaccine decreases recurrent virus shedding and recurrent genital herpes disease. Vaccine. 2019 Jun 6;37(26):3443-3450. doi: 10.1016/j.vaccine.2019.05.009. Epub 2019 May 15. PMID 31103365